CLINICAL TRIAL: NCT00868842
Title: Open-label, Single-center Study of Whether Oral Penicillin Desensitization of Healthy Sensitive Subjects Results in Allergen Cross-desensitization of Mast Cells by Skin Testing and Desensitization of Peripheral Blood Basophils.
Brief Title: Desensitization of Human Mast Cells: Mechanisms and Potential Utility for Preventing Anaphylaxis
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: HM10870; AADCRC-VCU-01
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Anaphylaxis
Keywords: Penicillin; Allergy; Prevention; Anaphylaxis; Clinically proven history of penicillin allergy; preventing anaphylaxis
MeSH Terms: conditions — Anaphylaxis; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an open-label, single-center study of whether oral penicillin desensitization of healthy sensitive subjects results in allergen cross-desensitization of mast cells by skin testing and desensitization of peripheral blood basophils. The primary endpoint(s) will be PC3 prick skin test values to penicillin, aeroallergen(s) and codeine. Secondary endpoints will be levels of Syk in purified basophils determined by flow cytometry (mean fluorescence intensity) and basophil degranulation (% tryptase release) to anti-FcåRI and to calcium ionophore.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Male, or non-pregnant female, 18-45 years of age who are in good health.
* Clinical history of a penicillin allergy consisting of an immediate hyper- sensitivity reaction such as anaphylaxis, urticaria/angioedema or broncho- spasm, and a positive skin prick test to penicillin G.
* Positive skin test to at least one aeroallergen to indicate sensitivity, but clinical disease (allergic rhinitis) is not necessary.

Exclusion Criteria:

* Dermatographism or severe dermatologic condition, such as advanced eczema or psoriasis, that will not allow an adequate uninvolved area for skin testing.
* Negative skin tests to penicillin G or to all aeroallergens test.
* Pregnancy.
* Antihistamine medications taken within one week of testing; systemic steroids, B-blockers or ACE -inhibitors taken over the previous month; omalizumab therapy at any time; those receiving or who have received immunotherapy; and those who have been desensitized to any drug within 6 months.
* Allergic reaction to a B-lactam antibiotic within 1 month.
* Current asthma; significant pulmonary, cardiovascular, renal, hepatobiliary or neurological diseases, or another disease process that the investigator feel would put the subject at risk of an adverse event.
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
* Inability or unwillingness of a participant to give written informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Clinical and community recruitment
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Decreased skin test sensitivity to Pre-pen (PC3 value) | June 2012

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence B. Schwartz, M.D., Ph.D, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States